CLINICAL TRIAL: NCT02414971
Title: Relationship of Mitochondrial Enzymes With Cancer Related Fatigue
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201500023-N; OCR14952 (Other: University of Florida); pending (Other: National Institute of Nursing Research)
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Prostate Cancer
Keywords: cancer related fatigue; prostate cancer; mitochondria
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Buccal swabs Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men with prostate cancer: men over 18 years of age diagnosed with prostate cancer receiving external beam radiation
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
Project Study: Pilot Human Study Specific Aims: 1. describe levels of mitochondrial respiratory enzymes 2. examine relationships between levels of mitochondrial enzymes, fatigue, and health-related quality of life; and 3. compare levels of mitochondrial enzymes in men with a clinically-significant change in fatigue from those with no change in fatigue.

Significance of Study: Cancer related fatigue is a common side effect of cancer. Cancer related fatigue is poorly understood. Many different biological mechanisms have been theorized, including mitochondrial dysfunction. Self-reported descriptions of reduced energy and muscle weakness lend support for a possible relationship of cancer related fatigue to mitochondrial dysfunction.

Main Research Variables: Mitochondrial Enzymes, Cancer related fatigue, and health related quality of life Design: Descriptive, longitudinal study Sample/Setting: Men with non-metastatic prostate-cancer who are scheduled to receive radiation therapy Methods: Questionnaires, mouth swabs and blood will be collected at four study visits: prior to treatment, midpoint of treatment, completion of treatment and within 90 days of finishing treatment. Four mouth swabs will be collected per participant at each study visit.

Implications for Practice: Understanding the role of mitochondrial enzymes in cancer related fatigue has major clinical implications in the development of targeted interventions and in providing specific knowledge for patients and their families to make informed treatment decisions.

DETAILED DESCRIPTION:
Project Narrative

Purpose and Specific Aims The primary purpose of this pilot study is to explore the relationship between mitochondria and fatigue in men diagnosed prostate cancer. The specific aims are to: (a) describe levels of mitochondrial enzymes, (b) examine relationships between levels of mitochondrial enzymes, fatigue, and health-related quality of life (HRQOL); and (c) compare levels of mitochondrial enzymes in men with and without fatigue.

Methods Design The proposed study will use a descriptive, longitudinal design to describe levels of mitochondrial enzymes Sample and Setting Men with prostate cancer who are scheduled to receive radiation at the University of Florida Health Cancer Center will be eligible for study participation. Men will be enrolled if they: (a) have prostate cancer (b) are scheduled to receive radiation and (c) are at least 18 years of age. Patients will be excluded if they: (a) have any inflammatory or infectious condition such as rheumatoid arthritis, lupus, or cirrhosis; an infectious disease such as HIV, tuberculosis, or hepatitis; (b) have other types of cancer; (c) had a major psychiatric disorder or alcohol or drug abuse within the past 5 years; (d) are receiving or scheduled to receive chemotherapy; or (e) are taking steroids, non-steroidal anti-inflammatories, or tranquilizers.

Experimental Variables:

The primary purpose of this study is to describe levels of mitochondrial enzymes, Cancer related fatigue and health related quality of life.

All mouth swab samples collected will be coded and stored in a secured freezer. The frozen buccal swab samples will be batch shipped to the National Institute of Nursing Research and then processed and shipped to St. Christopher's Hospital for Children of Philadelphia for analyses.

Data Collection Schedule Study time points. Data will be collected at four study visits: baseline, midpoint of treatment, completion of treatment and within 90 days after treatment. Four buccal swabs will be collected per participant at each study visit using the Epicentre Catch-All Sample Collection Swabs-Soft Pack.

Study Procedures. The patients included in this study will be consented and enrolled into an Institutional Review Board-approved protocol for men with prostate cancer who are scheduled to receive radiation treatment. Biologic (buccal swabs) and questionnaire (Functional Assessment of Cancer Therapy-Prostate) data will be collected at each of four study visits. Each study visit will be arranged to coincide with scheduled clinic visits to decrease patient burden.

ELIGIBILITY:
Inclusion Criteria: diagnosis of prostate cancer, non metastatic, over 18 years of age, scheduled to receive external beam radiation, -

Exclusion Criteria: have any inflammatory or infectious condition such as rheumatoid arthritis, lupus, or cirrhosis; an infectious disease such as HIV, tuberculosis, or hepatitis; have other types of cancer; had a major psychiatric disorder or alcohol or drug abuse within the past 5 years; (d) are receiving or scheduled to receive chemotherapy; or are on a prescribed anti-inflammatory regimen such as steroids, non-steroidal anti-inflammatories, or tranquilizers.

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men over 18 years of age diagnosed with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-Prostate (FACT-P) | up to 180 days after completion of radiation
  The FACT-P is a 39 item scale with a range of 0-140. Higher scores mean higher health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Debra L Kelly, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States